CLINICAL TRIAL: NCT01271257
Title: Phase 1 Study of Titrated Oral Misoprostol
Brief Title: Pharmacokinetics of Misoprostol With Titrated Oral Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Shi-Yann Cheng, Director of Department of Obstetrics and Gynecology, China Medical University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CMUBH R990011; DMR-IRB-242 (Other: China Medical University Hospital)
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Hypotonic; Labor
Keywords: misoprostol, pharmacokinetics
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hourly misoprostol (Experimental): 20 microgram misoprostol intake per hour
  Interventions: Drug: Misoprostol
- traditional misoprostol (Active Comparator): 80 microgram misoprostol intake per 4 hours
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — 20 microgram PO per hour for 8 doses or 80 microgram PO per 4 hours for 2 doses
  Other Names: cytotec

SUMMARY:
The AUC240, AUC360, and AUC480 of titrated oral misoprostol are greater than traditional oral misoprostol.

DETAILED DESCRIPTION:
The primary outcomes measures of the study are the area under the curve of serum concentration of misoprostol acid against time up to 240, 360 and 480 minutes.

ELIGIBILITY:
Inclusion Criteria:

* 20-40 Y/O healthy and non-pregnant woman

Exclusion Criteria:

* heart, liver or kidney disease, anaphylaxis to misoprostol

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
AUC480 (the area under the curve of serum concentration of misoprostol acid against time up to 480 minutes) | 480 min post start of oral misoprostol administration

SECONDARY OUTCOMES:
AUC240 (the area under the curve of serum concentration of misoprostol acid against time up to 240 minutes) | 240 min post start of oral misoprostol administration
AUC360 (the area under the curve of serum concentration of misoprostol acid against time up to 360 minutes) | 360 min post start of oral misoprostol administration

CONTACTS AND LOCATIONS:
Overall Officials: Shi-Yann Cheng, M.D., Principal Investigator — China Medical University Beigang Hospital
Locations (1):
- China Medical University Beigang Hospital, Yunlin Xian, Taiwan, Taiwan

REFERENCES:
- [Background] Tang OS, Schweer H, Seyberth HW, Lee SW, Ho PC. Pharmacokinetics of different routes of administration of misoprostol. Hum Reprod. 2002 Feb;17(2):332-6. doi: 10.1093/humrep/17.2.332. PMID 11821273
- [Background] Zieman M, Fong SK, Benowitz NL, Banskter D, Darney PD. Absorption kinetics of misoprostol with oral or vaginal administration. Obstet Gynecol. 1997 Jul;90(1):88-92. doi: 10.1016/S0029-7844(97)00111-7. PMID 9207820
- See also: China Medical University Beigang Hospital — http://www.bh.cmu.edu.tw/cmubh/ch/index.php